CLINICAL TRIAL: NCT03330132
Title: Immunogenicity of Alternative Annual Influenza Vaccination Strategies in Older Adults in Hong Kong - a Randomized Controlled Trial
Brief Title: Immunogenicity of Alternative Annual Influenza Vaccination Strategies in Older Adults in Hong Kong
Acronym: PIVOT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YHT005.1
Record Dates: First submitted 2017-10-10; First posted 2017-11-06 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Annual vaccination with standard influenza vaccine or enhanced influenza vaccine, including some combination strategies (alternating each year) and some strategies with the same vaccine administered each year
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Standard vaccine (Active Comparator): Once-annual administration of standard vaccine (northern hemisphere formulation) prior to the northern hemisphere winter throughout 4 years study period.
  Interventions: Biological: Standard inactivated influenza vaccine (NH formulation)
- Alternating standard vaccine & adjuvanted vaccine (Experimental): Alternating once-annual administration of standard inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter, and once-annual administration of MF59 adjuvanted inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter throughout 4 years study period.
  Interventions: Biological: Standard inactivated influenza vaccine (NH formulation); Biological: MF 59 adjuvanted inactivated influenza vaccine (NH formulation)
- Alternating adjuvanted vaccine & standard vaccine (Experimental): Alternating once-annual administration of MF59 adjuvanted inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter, and once-annual administration of standard inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter throughout 4 years study period.
  Interventions: Biological: Standard inactivated influenza vaccine (NH formulation); Biological: MF 59 adjuvanted inactivated influenza vaccine (NH formulation)
- Alternating standard vaccine and high-dose vaccine (Experimental): Alternating once-annual administration of standard inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter, and once-annual administration of high-dose inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter throughout 4 years study period.
  Interventions: Biological: Standard inactivated influenza vaccine (NH formulation); Biological: High-dose inactivated influenza vaccine (NH formulation)
- Alternating high-dose vaccine and standard vaccine (Experimental): Alternating once-annual administration of high-dose inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter, and once-annual administration of standard inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter throughout 4 years study period.
  Interventions: Biological: Standard inactivated influenza vaccine (NH formulation); Biological: High-dose inactivated influenza vaccine (NH formulation)
- Alternating adjuvanted vaccine and high-dose vaccine (Experimental): Alternating once-annual administration of MF59 adjuvanted inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter, and once-annual administration of high-dose inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter throughout 4 years study period.
  Interventions: Biological: MF 59 adjuvanted inactivated influenza vaccine (NH formulation); Biological: High-dose inactivated influenza vaccine (NH formulation)
- Alternating high-dose vaccine and adjuvanted vaccine (Experimental): Alternating once-annual administration of high-dose inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter, and once-annual administration of MF59 adjuvanted inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter throughout 4 years study period.
  Interventions: Biological: MF 59 adjuvanted inactivated influenza vaccine (NH formulation); Biological: High-dose inactivated influenza vaccine (NH formulation)
- High-dose vaccine (Experimental): Once-annual administration of high-dose inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter throughout 4 years study period.
  Interventions: Biological: High-dose inactivated influenza vaccine (NH formulation)
- Adjuvanted vaccine (Experimental): Once-annual administration of MF59 adjuvanted inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter throughout 4 years study period.
  Interventions: Biological: MF 59 adjuvanted inactivated influenza vaccine (NH formulation)
- Recombinant vaccine (Experimental): Once-annual administration of recombinant hemagglutinin inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter throughout 4 years study period.
  Interventions: Biological: Recombinant hemagglutinin inactivated influenza vaccine (NH formulation)
- Alternating recombinant vaccine and adjuvanted vaccine (Experimental): Alternating once-annual administration of recombinant hemagglutinin inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter, and once-annual administration of MF59 adjuvanted inactivated influenza vaccine (northern hemisphere formulation) prior to the northern hemisphere winter throughout 4 years study period.
  Interventions: Biological: MF 59 adjuvanted inactivated influenza vaccine (NH formulation); Biological: Recombinant hemagglutinin inactivated influenza vaccine (NH formulation)

INTERVENTIONS:
Biological: Standard inactivated influenza vaccine (NH formulation) — 0.5mL FluQuadri®, Sanofi Pasteur, containing 60μg antigen - 15μg for each influenza strain included - with strains recommended by the WHO for the northern hemisphere formulation.
  Arms: Alternating adjuvanted vaccine & standard vaccine; Alternating high-dose vaccine and standard vaccine; Alternating standard vaccine & adjuvanted vaccine; Alternating standard vaccine and high-dose vaccine; Standard vaccine
Biological: MF 59 adjuvanted inactivated influenza vaccine (NH formulation) — 0.5mL FLUAD(TM), Seqirus containing 45μg antigen; 15μg for each influenza strain included and MF59C.1 adjuvant (MF59®) with strains recommended by the WHO for the northern hemisphere formulation.
  Arms: Adjuvanted vaccine; Alternating adjuvanted vaccine & standard vaccine; Alternating adjuvanted vaccine and high-dose vaccine; Alternating high-dose vaccine and adjuvanted vaccine; Alternating recombinant vaccine and adjuvanted vaccine; Alternating standard vaccine & adjuvanted vaccine
Biological: High-dose inactivated influenza vaccine (NH formulation) — 0.5mL Fluzone® High-Dose, Sanofi Pasteur containing 180μg antigen; 60μg for each influenza strain included with strains recommended by the WHO for the northern hemisphere formulation.
  Arms: Alternating adjuvanted vaccine and high-dose vaccine; Alternating high-dose vaccine and adjuvanted vaccine; Alternating high-dose vaccine and standard vaccine; Alternating standard vaccine and high-dose vaccine; High-dose vaccine
Biological: Recombinant hemagglutinin inactivated influenza vaccine (NH formulation) — 0.5mL Flublok®, Protein Sciences Corporation containing 180μg antigen, 45μg for each influenza strain included with strains recommended by the WHO for the northern hemisphere formulation.
  Arms: Alternating recombinant vaccine and adjuvanted vaccine; Recombinant vaccine

SUMMARY:
This study allows to evaluate the strength and duration of immune responses between annual receipt of standard inactivated vaccine and alternative potent vaccines, including annual receipt of adjuvanted inactivated vaccine, annual receipt of high-dose inactivated vaccine, annual receipt of recombinant HA vaccine, and the alternate combinations of the former three vaccines over four years, for identifying improved vaccination strategies for influenza vaccination in older adults in a location experiencing a subtropical pattern in influenza activity.

DETAILED DESCRIPTION:
Background: The typical vaccination strategy of annual administration with inactivated trivalent influenza vaccine (TIV) or quadrivalent influenza vaccine (QIV) may provide suboptimal protection to older adults in a location with prolonged periods of influenza activity because of the weaker immune response of older adults to vaccination and because of post-vaccination waning in protection over the course of a year. We hypothesize that in a subtropical or tropical location with prolonged circulation of influenza viruses, the higher antibody titers over years achieved after receipt of annual high-dose vaccine, MF59-adjuvanted vaccine or recombinant haemagglutinin (HA) vaccine, or different vaccination strategies of their combinations with or without the standard vaccine, might lead to greater protection than annual receipt of standard vaccines.

Aim: To test the immune profiles over time of older adults following different influenza vaccination strategies.

Design and subjects: Initially a 4-year immunogenicity study with a randomized controlled design among 2200 older adults aged 65-82 years. We will enroll participants who are willing to receive annual influenza vaccination from the general community including community centres and day-care centres. Eligible individuals will be randomly allocated to ten intervention groups (i.e. annual standard QIV, annual MF59-adjuvanted TIV, annual high-dose TIV, annual recombinant-HA QIV, and six combinations of their alternate annual use) consisting of four rounds of vaccination before each winter influenza season and followed up for 4 years. For each round of vaccination, blood samples for immunological tests will be collected before vaccination and 30 and 182 days after vaccination in all participants, and also at 7, 91 and 273 days after vaccination in a subset of 10% of the participants. Acute illnesses among participants will be monitored by active surveillance efforts during influenza seasons. The vaccine formulation in each round of vaccination will be updated for each season according to WHO recommendations.

Study extension: In years 5-8, all participants will receive the recombinant-HA QIV once per year before each winter influenza season, and their receipt of COVID-19 vaccines will also be recorded. Samples will be collected at the same timepoints to monitor immune responses to influenza vaccination and how responses are affected by prior vaccination history.

Main outcome measures: Antibody titers measured by haemagglutination-inhibition assays, which is an established correlate of protection, in addition to other measurements on humoral and cell-mediated immune responses in the ten intervention groups each year.

ELIGIBILITY:
Inclusion Criteria:

• Adult aged 65-82 years attending ECC and EDC who has not received 2017/18 seasonal influenza vaccine and is willing to receive annual influenza vaccination

Exclusion Criteria:

* Individuals who show signs of dementia (do not pass the Mini-cog test under Appendix 1a: Recruitment Screening Log) or significant cognitive impairment and are not competent to give their consent.
* Individuals who report medical conditions not suitable to receive inactivated influenza vaccines, such as:

  * Severe allergic reaction (e.g., anaphylaxis) after previous dose of any influenza vaccine; or to a vaccine component, including egg protein;
  * Moderate or severe acute illness with or without fever after any previous influenza vaccination; or
  * A history of Guillain-Barré syndrome (GBS) within 6 weeks of previous influenza vaccination.
* Individuals, who report medical conditions not suitable to receive intramuscular injection, such as:

  * bleeding disorders
  * habitually taking anticoagulants (with the exception of antiplatelets such as aspirin).
* Individuals who have any medical conditions not suitable to receive inactivated influenza vaccines as determined by a clinician.

Ages: 65 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1861 (Actual)
Dates: Start 2017-10-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference in antibody titres | 30 and 182 days after each vaccination
  The difference in antibody titres of participants measured by haemagglutination-inhibition (HAI) assay, evaluated by (1) the proportion of participants who achieve a target rise in antibody titre against each of the vaccine strains at 30 days, and (2) the geometric mean titre (GMT) ratios between the two groups against each of the vaccine strains at 30 days and 182 days. (The targeted rise in antibody titre is defined as the percentage of subjects with either a pre-vaccination HAI titre <10 and a post-vaccination HAI titre ≥40, or a pre-vaccination HAI titre ≥10 and a minimum four-fold rise in post-vaccination HAI antibody titre.)

SECONDARY OUTCOMES:
Seroprotection | 30 days after each vaccination
  The proportion of participants who achieve seroprotection defined as an HAI titre ≥40 after each vaccination before the winter seasons.
CMI responses | . 7 days after each vaccination
  The vaccine-induced influenza-specific CD4+ and CD8+ T cell responses 7 days post- vaccination, proxy by anti-viral IFNγ production evaluated by Intracellular Cytokine Staining (ICS) assay. Responses for these and other relevant biomarkers are compared to baseline at the time of vaccination.
Adverse events | 30 days after each vaccination
  The rate of adverse events within 30 days after vaccination for each round of vaccination.
PCR confirmed infection | 182 days after each vaccination
  The rate of PCR-confirmed influenza infection in each round of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J COWLING, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Fox A, Sanchez-Ovando S, Carolan L, Hadiprodjo AJ, Chen Y, Ho F, Cheng SMS, Thompson MG, Iuliano AD, Levine MZ, Valkenburg SA, Ip DKM, Peiris JSM, Sullivan SG, Cowling BJ, Leung NHL. Enhanced Influenza Vaccines Extend A(H3N2) Antibody Reactivity in Older Adults but Prior Vaccination Effects Persist. Clin Infect Dis. 2025 Nov 6;81(4):e192-e201. doi: 10.1093/cid/ciaf060. PMID 40178253
- [Derived] Cowling BJ, Thompson MG, Ng TWY, Fang VJ, Perera RAPM, Leung NHL, Chen Y, So HC, Ip DKM, Iuliano AD. Comparative Reactogenicity of Enhanced Influenza Vaccines in Older Adults. J Infect Dis. 2020 Sep 14;222(8):1383-1391. doi: 10.1093/infdis/jiaa255. PMID 32407535
- [Derived] Cowling BJ, Perera RAPM, Valkenburg SA, Leung NHL, Iuliano AD, Tam YH, Wong JHF, Fang VJ, Li APY, So HC, Ip DKM, Azziz-Baumgartner E, Fry AM, Levine MZ, Gangappa S, Sambhara S, Barr IG, Skowronski DM, Peiris JSM, Thompson MG. Comparative Immunogenicity of Several Enhanced Influenza Vaccine Options for Older Adults: A Randomized, Controlled Trial. Clin Infect Dis. 2020 Oct 23;71(7):1704-1714. doi: 10.1093/cid/ciz1034. PMID 31828291